CLINICAL TRIAL: NCT05727865
Title: Online Cognitive Behavioral Therapy for Rehabilitation After Cardiac Surgery
Acronym: TRACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Josefin Särnholm, PhD, Lic. Psychologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRACS-PILOT
Record Dates: First submitted 2023-02-06; First posted 2023-02-14 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Surgery
Keywords: Psychological distress; Cognitive behavioral therapy; Fatigue; Depression; Anxiety
MeSH Terms: conditions — Fatigue; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online CBT following cardiac surgery (Experimental): The treatment lasts for five weeks and will be provided as an early intervention following cardiac surgery ≥ eight weeks to nine months before assessment. The intervention is psychologist-guided (clinical psychologist and/or resident psychologist under supervision) and delivered via text-based interactive online treatment modules, where patients complete weekly homework assignments and have regular online contact with psychologists with training in CBT for cardiac disease.
  Interventions: Behavioral: Online CBT following cardiac surgery

INTERVENTIONS:
Behavioral: Online CBT following cardiac surgery — It will include psychoeducation, behavioral activation to address post-operative fatigue and depression, interoceptive exposure to reduce fear of cardiac-related symptoms and in-vivo exposure to reduce avoided situations, and activities to enhance physical activity and wellbeing. Labeling (i.e., describing post-operative and/or cardiac-related symptoms, thoughts, and feelings) will be used continuously during treatment to enhance the effect of exposure and pain management

SUMMARY:
The purpose of the present pilot study is to evaluate the feasibility and potential efficacy of a brief, internet-delivered CBT protocol provided early following cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery is a major surgical procedure used to treat for example coronary artery disease (CAD). The intervention increases survival rates and reduces cardiac symptom burden in cardiac patients. However, cardiac surgery is associated with elevated symptoms of psychological distress, which are related to several negative outcomes, such as poorer health-related quality of life (QoL) and response to treatment. There is a clear need to develop a brief psychological intervention that can be provided early in the clinical course after cardiac surgery to reduce psychological distress.

The purpose of this pilot study is to evaluate the feasibility and potential efficacy of a brief, exposure-based internet-delivered CBT protocol provided early after cardiac surgery. This is an uncontrolled pilot study with a pretest-posttest design. The study will include 30 participants. Assessments will be conducted pre-treatment, post-treatment, one- and six months after treatment. The one-month follow-up is the primary endpoint.

The treatment lasts for five weeks and will be provided as an early intervention following cardiac surgery ≥ eight weeks to nine months before assessment. It will include psychoeducation, behavioral activation to address post-operative fatigue and depression, interoceptive exposure to reduce fear of cardiac-related symptoms and in-vivo exposure to reduce avoided situations, and activities to enhance physical activity and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* (A) Cardiac surgery (i.e., CABG, heart valve repair/replacement, aortic repair or combined CABG and valve repair/replacement) ≥ eight weeks to nine months before assessment
* (B) Age 18 years and above;
* (C) Endorses postoperative psychological distress and/or interference with daily life
* (D) On medical treatment for the cardiac condition according to clinical guidelines;
* (E) Ability to read and write in Swedish

Exclusion Criteria:

* (F) Prior cardiac surgery with ventricular assist device or heart transplant;
* (G) Hospitalized or living in a care facility;
* (H) Any medical restriction to be physical active;
* (I) Severe medical illness i.e., terminal cancer ;
* (J) Severe psychiatric disorder or risk of suicide;
* (K) Alcohol dependency;
* (L) Ongoing psychological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
12-Item Short-Form Health Survey | Baseline to 2 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
Acceptability: Client satisfaction Questionnaire | Baseline to 5 weeks.
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
Percentage of enrolled participants who complete the treatment | Baseline to 5 weeks
  Feasibility of the intervention components will be assessed by >60% assessed as treatment completers. Descriptive analysis will also provide number of messages and therapist time.
Adverse events | Baseline to 5 weeks
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').

SECONDARY OUTCOMES:
12-Item Short-Form Health Survey | Baseline to 5 weeks
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
12-Item Short-Form Health Survey | Baseline to 7 months
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life
Cardiac anxiety questionnaire | Baseline to 5 weeks
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | Baseline to 2 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | Baseline to 7 months
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Patient Health Questionnaire-9 | Baseline to 5 weeks
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | Baseline to 2 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Patient Health Questionnaire-9 | Baseline to 7 months
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression
Generalized Anxiety Disorder 7-item | Baseline to 5 weeks
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | Baseline to 2 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | Baseline to 7 months
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Brief Pain Inventory Short Form | Baseline to 5 weeks
  Measure of pain interference and severity, with a higher score indicating more pain.
Brief Pain Inventory Short Form | Baseline to 2 months
  Measure of pain interference and severity, with a higher score indicating more pain.
Brief Pain Inventory Short Form | Baseline to 7 months
  Measure of pain interference and severity, with a higher score indicating more pain.
Multidimensional fatigue inventory | Baseline to 5 weeks
  Measure of fatigue, with a higher score indicating more fatigue.
Multidimensional fatigue inventory | Baseline to 2 months
  Measure of fatigue, with a higher score indicating more fatigue.
Multidimensional fatigue inventory | Baseline to 7 months
  Measure of fatigue, with a higher score indicating more fatigue.
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | Baseline to 5 weeks
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | Baseline to 2 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
Symptom checklist Severity and Frequency Scale (SCL, adapted to coronary artery disease) | Baseline to 7 months
  Cardiac-related symptoms in two sub scales A) frequency: score ranging from 0-48, with higher score indicating higher frequency of symptoms, B) severity of experienced symptom: score ranging from 0- 48, with a higher score indicating more severe symptoms
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to weeks
  evel of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 2 months
  evel of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
The Godin Leisure-time Exercise and International Physical Activity Questionnaire 1 item on inactivity | Baseline to 7 months
  evel of physical activity and inactivity: On the Godin leisure-time excercise: The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity. And from International Physical Activity Questionnaire we will use 1 item on inactivity
University of Toronto Atrial fibrillation Severity Scale (AFSS) | Baseline to 5 weeks
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | Baseline to 2 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.
University of Toronto Atrial fibrillation Severity Scale (AFSS) | Baseline to 7 months
  3 item on cardiac-specific healthcare consumption. Scores ranges 0-15 with a higher score indicating more cardiac-related healthcare consumption.

OTHER OUTCOMES:
Adverse events | Baseline to 2 months
  otential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | Baseline to 7 months
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').

CONTACTS AND LOCATIONS:
Overall Officials: Josefin Särnholm, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden